CLINICAL TRIAL: NCT04135820
Title: An Open-label, Randomised, Single Dose, Cross-over Phase I Study to Determine the Effect of Food on the Pharmacokinetic Profile of BPI-7711
Brief Title: A Phase I Study to Determine the Effect of Food on the Pharmacokinetic Profile of BPI-7711
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beta Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BPI-7711FE
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: NSCLC
MeSH Terms: interventions — rezivertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasted (Experimental): BPI-7711 following a period of fasting
  Interventions: Drug: BPI-7711
- High-fat meal (Experimental): BPI-7711 following a high-fat meal.
  Interventions: Drug: BPI-7711

INTERVENTIONS:
Drug: BPI-7711 — BPI-7711 180 mg
  Other Names: BPI-7711 capsule

SUMMARY:
This is an open-label, randomised, single-dose, cross-over phase I study to evaluate the effect of food on the pharmacokinetic profile of BPI-7711 in Chinese healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged from 18 to 55 years.
* BMI from 18.5 to 28.0 kg/m2
* Medical history, vital signs, physical examination and lab tests are normal or abnormal without clinical significance.

Exclusion Criteria:

* Subjects with clinical significant diseases
* Subjects with allergic disease history
* Subjects with gastrointestinal disease history that can affect study drug absorption
* Subjects with drug abuse history

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Cmax | Blood samples collected on Day 1 and Day 15 at pre-dose, 1, 2, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144 and 168 hours post BPI-7711 dose
  Pharmacokinetics of BPI-7711 by assessment of maximum plasma concentration
AUC(0-last) | Blood samples collected on Day 1 and Day 15 at pre-dose, 1, 2, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144 and 168 hours post BPI-7711 dose
  Pharmacokinetics of BPI-7711 by assessment of area under the plasma concentration time curve from zero to last assessed timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Yongfang Yuan, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No